CLINICAL TRIAL: NCT04736303
Title: Assessing the Impact of the Implementation of BIS on the Incidence of Postoperative Delirium - A Monocentre Prospective Trial
Brief Title: The Impact of the Implementation of BIS on the Incidence of Postoperative Delirium
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Elena Arnaoutoglou, Professor of Anesthesiology, University of Thessaly
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: POD and BIS
Record Dates: First submitted 2020-10-02; First posted 2021-02-03 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POD without BIS (No Intervention): Assessing the incidence of POD in patients under general anethesia for elective non cardiac surgery, with CAM and Nu-DESC tools.
- POD with BIS (Active Comparator): Assessing the incidence of POD in patients under general anethesia for elective non cardiac surgery with the implementation of BIS monitoring, with CAM and Nu-DESC tools.
  Interventions: Device: BIS

INTERVENTIONS:
Device: BIS — The implementation of BIS monitoring
  Arms: POD with BIS

SUMMARY:
This study will investigate the incidence of postoperative POD in patients undergoing non cardiac surgery under general anesthesia with and without the implementation of the BIS monitoring.T

DETAILED DESCRIPTION:
This study will compare the incidence of POD after elective non cardiac surgery conducted under general anesthesia before and after the implementation of BIS monitoring in our University Hospital.

The POD will be evaluated with the CAM and Nu-DESC tools, which have been adapted for the greek population.

ELIGIBILITY:
Inclusion Criteria:

1. adult patients over 60 years of age
2. an American Society of Anesthesiologists (ASA) physical status I to III
3. undergoing elective non cardiac surgery under general anaesthesia
4. native speakers of the Greek language
5. eligible to leave the post-anaesthesia care unit
6. an expected in-hospital stay at least 24 hours following surgery

Exclusion Criteria:

1. refused to participate or sign the informed consent form
2. surgery or anaesthesia within the last 30 day
3. any prior or current history involving an affliction of the central nervous system
4. severe hearing or visual impairment
5. psychiatric disorders
6. a score less than 5 according the Geriatric Depression Scale (GDS-15)
7. a score less than 4 for females and less than 2 for males according to the Lawton-Brody Instrumental Activities of Daily Living Scale (I.A.D.L.)
8. alcohol consumption less than 35 units/week
9. drug dependence
10. previous neuropsychological testing
11. haemodynamical instability
12. peri-procedural desaturation (one or more events of SpO2<80% for more than 2 minutes)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of POD | 1st postoperative day
  Assess the incidence of POD with CAM and Nu-DESC tools

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Arnaoutoglou, MD, PhD, Study Chair — University of Thessaly; Maria Ntalouka, MD, PhD, Principal Investigator — University Hospital of Larissa
Locations (1):
- Univeristy of Thessaly, Larissa, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: Undecided